CLINICAL TRIAL: NCT05469152
Title: Accuracy of Detachable String Magnetically Controlled Capsule Endoscopy for Follow-up of Patients With Esophageal Diseases: A Multicenter Study
Brief Title: Detachable String Magnetically Controlled Capsule Endoscopy for Follow-up of Patients With Esophageal Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Ruijin Hospital (Other); Shanghai Zhongshan Hospital (Other); XuHui District Central Hospital (Unknown); Yangpu District Central Hospital Affiliated to Tongji University (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Professor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DS-MCE-esophagus
Record Dates: First submitted 2022-07-11; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Esophageal Diseases
Keywords: esophageal diseases; capsule endoscopy
MeSH Terms: conditions — Esophageal Diseases | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ds-MCE and EGD (Experimental): All the enrolled participants will undergo the examination of detachable string magnetically controlled capsule endoscopy (ds-MCE) first, followed by EGD within 48 hours.
  Interventions: Diagnostic Test: ds-MCE and EGD

INTERVENTIONS:
Diagnostic Test: ds-MCE and EGD — Procedure of ds-MCE: The ds-MCE system mainly consists of two parts: the NaviCam magnetic capsule endoscopy guidance system and the detachable string part. The capsule, which is partially enclosed within the sleeve, can be actively moved in the esophagus through the control of string. Investigator can examine the entire esophagus several times under real time views. The capsule then could be detached from the string system through injecting air into the hollow string with the syringe after completing the examination of esophagus. Then, the examination of stomach under magnetic control and small bowel under the natural action of peristalsis follows.
  Procedure of EGD: The EGD will be performed using conventional upper gastrointestinal video endoscopy, according to the standard procedure at individual centers. EGD will be performed within 48 hours after ds-MCE procedure and usually during the same endoscopic session.

SUMMARY:
The purpose of the study is to determine the accuracy of detachable string magnetically controlled capsule endoscopy(DS-MCE) as a follow-up method for patients with previous esophageal diseases.

DETAILED DESCRIPTION:
Esophagogastroduodenoscopy (EGD) is recognized as the gold standard for detection and follow-up of esophageal diseases,allowing for direct mucosal visualization and therapeutic intervention. EGD is however an invasive procedure and there is potential for procedure-related complications, such as perforation and bleeding.Esophageal capsule endoscopy(ECE)provides a novel noninvasive approach to visualize the esophagus.The main drawback for the use of ECE is its unreliable transit time which often renders an inadequate visualization of the esophagus.Thus investigators have developed the detachable string magnetically controlled capsule endoscopy(DS-MCE) which can control the movement of the capsule through the string.

The ds-MCE system consists of two parts: the magnetically controlled capsule endoscopy (MCE) system and a transparent latex sleeve with a hollow string. The magnetically controlled capsule endoscopy (MCE) system (Ankon Technologies, Shanghai, China) detects focal lesions in the stomach with comparable accuracy with conventional EGD. One end of the hollow string is a transparent thin latex sleeve that can be wrapped on the surface of the capsule, and the other end of the string is connected to the syringe. The capsule, which is partially enclosed within the sleeve, can be actively moved in the esophagus through the control of string. In this case, investigator can examine the entire esophageal mucosa several times under real time views. The capsule then could be detached from the string system through injecting air into the hollow string with the syringe after completing the examination of esophagus. The pilot study of ds-MCE confirmed it was a feasible, safe and well-tolerated method for completely viewing esophagus and stomach, without the need for sedation. Besides, the 8-10h battery life of the ds-MCE enables complete examination of the small bowel, which provides the possibility for screening pathological changes in the entire gastrointestinal tract.

This study is a prospective, multi-centered, diagnostic accuracy study. The primary outcome is the diagnostic accuracy of ds-MCE in identifying esophageal diseases. Second outcomes include the visualization and cleanliness of Z-line, safety and patient satisfaction of DS-MCE.

ELIGIBILITY:
Inclusion Criteria:

1. Gender is not limited.
2. Patients aged between 18-75 years or older.
3. Both inpatients and outpatients.
4. Patients with previous esophageal diseases who are scheduled to undergo EGD for follow-up.
5. Able to provide informed consent.

Exclusion Criteria:

1. Patients aged less than 18 years.
2. Patients with active upper gastrointestinal bleeding.
3. Patients who have participated in or are participating in other clinical trials within three months.
4. Patients with cancer on active treatment with chemotherapy and/or radiation therapy.
5. Pregnancy or suspected pregnancy.
6. Suspected or known intestinal stenosis or other known risk factors for capsule retention.
7. Pacemaker or other implanted electromedical devices which could interfere with magnetic resonance.
8. Patients with dysphagia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of the ds-MCE in identifying esophageal diseases in comparison to standardized EGD | 2 weeks
  To assess the diagnostic accuracy of the ds-MCE as a follow-up method for patients with previous esophageal diseases, using EGD as the gold standard.

SECONDARY OUTCOMES:
Number of quadrants visualized at Z-line by ds-MCE | 2 weeks
  To assess the visualization of Z-line. Circumferential visualization of the Z line by ds-MCE was defined by quadrants as follows: Z line not observed at all; less than 2 quadrants (< 50 %) of the Z line observed; between 2 quadrants and 3 quadrants (50 % - 75%) observed; more than 3 quadrants (> 75%) observed; and entire Z line (100 %) observed.
Scores of cleanliness of Z-line area | 2 weeks
  The effect of bubbles/saliva on the appearance of the Z line area was scored as follows: 0 = no interference by bubbles/saliva on the Z line area; 1 = minor interference of bubbles/saliva on the Z line area; 2 = major interference of bubbles/saliva on the Z line area.
Number of ds-MCE associated adverse events | 2 weeks
  To assess the safety of ds-MCE.
The patient satisfaction of the ds-MCE through questionnaires | 2 weeks
  To assess the patient satisfaction of the ds-MCE compared to standard EGD.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Principal Investigator — Changhai Hospital
Locations (7):
- China (7):
  - Ruijin Hospital, Shanghai
  - Shanghai Changhai Hospital, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - Xuhui District Central Hospital, Shanghai
  - Yangpu District Central Hospital, Shanghai
  - Zhongshan Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
After finishing this study, we will make the data available to other researchers:
  including study protocol, statistical analysis plan (SAP), informed consent form (ICF), clinical study report (CSR)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 years.
Access Criteria: The website of the journal where the results published, and ClinicalTrials.gov web site.

REFERENCES:
- [Background] Chen YZ, Pan J, Luo YY, Jiang X, Zou WB, Qian YY, Zhou W, Liu X, Li ZS, Liao Z. Detachable string magnetically controlled capsule endoscopy for complete viewing of the esophagus and stomach. Endoscopy. 2019 Apr;51(4):360-364. doi: 10.1055/a-0856-6845. Epub 2019 Mar 1. PMID 30822803
- [Background] de Franchis R, Eisen GM, Laine L, Fernandez-Urien I, Herrerias JM, Brown RD, Fisher L, Vargas HE, Vargo J, Thompson J, Eliakim R. Esophageal capsule endoscopy for screening and surveillance of esophageal varices in patients with portal hypertension. Hepatology. 2008 May;47(5):1595-603. doi: 10.1002/hep.22227. PMID 18435461
- [Background] Chen WS, Zhu LH, Li DZ, Chen L, Wu YL, Wang W. String esophageal capsule endoscopy with real-time viewing improves visualization of the distal esophageal Z-line: a prospective, comparative study. Eur J Gastroenterol Hepatol. 2014 Mar;26(3):309-12. doi: 10.1097/MEG.0000000000000038. PMID 24429971
- [Background] de Franchis R. Updating consensus in portal hypertension: report of the Baveno III Consensus Workshop on definitions, methodology and therapeutic strategies in portal hypertension. J Hepatol. 2000 Nov;33(5):846-52. doi: 10.1016/s0168-8278(00)80320-7. No abstract available. PMID 11097497
- [Background] Zou WB, Hou XH, Xin L, Liu J, Bo LM, Yu GY, Liao Z, Li ZS. Magnetic-controlled capsule endoscopy vs. gastroscopy for gastric diseases: a two-center self-controlled comparative trial. Endoscopy. 2015 Jun;47(6):525-8. doi: 10.1055/s-0034-1391123. Epub 2015 Jan 15. PMID 25590177
- [Background] Liao Z, Hou X, Lin-Hu EQ, Sheng JQ, Ge ZZ, Jiang B, Hou XH, Liu JY, Li Z, Huang QY, Zhao XJ, Li N, Gao YJ, Zhang Y, Zhou JQ, Wang XY, Liu J, Xie XP, Yang CM, Liu HL, Sun XT, Zou WB, Li ZS. Accuracy of Magnetically Controlled Capsule Endoscopy, Compared With Conventional Gastroscopy, in Detection of Gastric Diseases. Clin Gastroenterol Hepatol. 2016 Sep;14(9):1266-1273.e1. doi: 10.1016/j.cgh.2016.05.013. Epub 2016 May 20. PMID 27211503
- [Background] Liao Z, Gao R, Xu C, Xu DF, Li ZS. Sleeve string capsule endoscopy for real-time viewing of the esophagus: a pilot study (with video). Gastrointest Endosc. 2009 Aug;70(2):201-9. doi: 10.1016/j.gie.2008.10.043. Epub 2009 Mar 14. PMID 19286182
- [Background] Hosoe N, Naganuma M, Ogata H. Current status of capsule endoscopy through a whole digestive tract. Dig Endosc. 2015 Jan;27(2):205-15. doi: 10.1111/den.12380. Epub 2014 Oct 20. PMID 25208463